CLINICAL TRIAL: NCT05485220
Title: The Effects of Arm Ergometer Endurance Training and High-intensity Interval Training on Respiratory Parameters, Musculoskeletal System, and Clinical Symptoms in Chronic Neck Pain
Brief Title: The Effects of Arm Ergometer Endurance Training and High-intensity Interval Training in Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sinem Ayyıldız Çinar, Principle Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-21111
Record Dates: First submitted 2022-02-20; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise; High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercise group (Experimental): the participants do aerobic training by an arm crank ergometer (Monark 881E Upper and Lower Body Ergometer)
  Interventions: Other: Aerobic exercise
- High intensity interval training group (Experimental): the participants do High intensity interval training by an arm crank ergometer (Monark 881E Upper and Lower Body Ergometer)
  Interventions: Other: High-intensity interval training
- control group (No Intervention): the participants don't do any exercises

INTERVENTIONS:
Other: Aerobic exercise — Aerobic exercise group: Peak workload will be determined by performing an exercise test on the patients. Training will be given at 60-70% of the peak workload for 45 minutes with an arm ergometer 3 days a week for 8 weeks.
  Arms: aerobic exercise group
Other: High-intensity interval training — High-intensity interval training Group: Peak workload will be determined by performing an exercise test on the patients and arm ergometer HIIT will be done with a total of 45 minutes, 90-95% of the peak workload for 30 seconds, 60 seconds in between, active recovery at 40-50% workload, 3 days a week for 8 weeks.
  Arms: High intensity interval training group

SUMMARY:
Neck pain is among the causes of morbidity that causes disability. Although it is not life-threatening, neck pain is one of the most important reasons for a decrease in the workforce. Since there is a close anatomical, musculoskeletal and neural connection between the cervical region and the thoracic spine, neck pain can affect respiratory functions by causing biomechanical changes in the thoracic spine and rib cage. The aim of this study is to investigate the effects of aerobic exercise and high-intensity interval training, which are known to have an effect on both the musculoskeletal system and respiratory functions, on the respiratory parameters and musculoskeletal system disorders and clinical outcomes of people with neck pain when applied with an arm ergometer.

DETAILED DESCRIPTION:
Patients will be divided into 3 groups as randomized controlled. Aerobic exercise will be applied to the first group and HIIT to the second group. The third group will be the control group.

The patients in the first group will be applied an aerobic exercise program with an arm ergometer. Peak workload will be determined by performing an exercise test with an arm ergometer and training will be given for 60-70% of the peak workload for 45 minutes with arm ergometer 3 days a week for 8 weeks.

HIIT with arm ergometer will be applied to the patients in the second group. Peak workload will be determined by performing an exercise test with an arm ergometer, and HIIT will be performed with an arm ergometer for 45 minutes in total, 90-95% of peak workload for 30 seconds, 60 seconds in between, active recovery at 40-50% workload. After the patients receive training for 8 weeks, 3 times a week, post-treatment evaluations will be made.

Only evaluations will be made twice, with an interval of 8 weeks, for the patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18-55,
* Having neck pain for more than 3 months,
* Having neck pain ≥3 cm in a 10 cm VAS and
* Patients with non-specific neck pain who score > 10/50 on the Neck Disability Index will be included.

Exclusion Criteria:

* Pregnant women,
* Smokers,
* BMI>40
* Those with any cardiovascular or pulmonary disease,
* Those who cannot exercise due to any medical condition,
* Those who have received physical therapy for neck pain in the last 6 months,
* Red flag (malignancy, spinal fracture, etc.),
* Spinal fracture,
* Shoulder fracture,
* Shoulder subluxation,
* Cervical or shoulder surgery,
* Migraine,
* Rheumatological diseases,
* Those with cervical root compression syndrome,
* Those with neurological/inflammatory spinal pathology,
* Those with chronic whiplash and traumatic neck injury,
* Persons with <24 points on the mini-mental test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
neck pain | 8 weeks
  participants' neck pain perception with visual analog pain scale. 0= no pain, 10=maximum pain
Spirometer measurements 1 | 8 weeks
  Forced Expiratory Volume during the first second (FEV1) with spirometer (Spirolab III, Spirolab, Medical International Research) (FEV1 and FVC will be combined to report FEV1/FVC)
Spirometer measurements 2 | 8 weeks
  Forced Vital Capacity (FVC) with spirometer (Spirolab III, Spirolab, Medical International Research) (FEV1 and FVC will be combined to report FEV1/FVC)
Spirometer measurements 3 | 8 weeks
  (FEV1/FVC) with spirometer (Spirolab III, Spirolab, Medical International Research) (FEV1 and FVC will be combined to report FEV1/FVC)
Spirometer measurements 4 | 8 weeks
  Forced Expiratory Flow (FEF%25-75) with spirometer (Spirolab III, Spirolab, Medical International Research)
MIP-MEP | 8 weeks
  maximal expiratory pressure (MEP) and maximal inspiratory pressure (MIP) with respiratory pressure meter (Micro Medical MicroMPM).
chest circumference measurement | 8 weeks
  chest circumference measurement with a tape measure.
Cervical Joint Range of Motion | 8 weeks
  Cervical Joint Range of Motion with Cervical Range of Motion - 3 (Performance Attainment Associates, St. Paul, MN, 55117, United States) (CROM 3).
Cervical Joint Position Error Test | 8 weeks
  Cervical Joint Position Error Test with Cervical Range of Motion - 3 (Performance Attainment Associates, St. Paul, MN, 55117, United States) (CROM 3).
Activation and endurance of deep cervical flexor muscles | 8 weeks
  Activation and endurance of deep cervical flexor muscles with Stabilizer Pressure Biofeedback.
craniovertebral angle | 8 weeks
  Craniovertebral angle will be measured by taking 2 lateral photographs of the subject. Spinous process of C7 and the tragus of ear will be marked with a body marker. A horizontal line is drawn passing through C7 making a right angle with the vertical. Then, the angle between the line connecting C7 spinous process with the tragus of the ear and the horizontal line, will measured using a goniometer
hand grip strength | 8 weeks
  Hand grip strength with Jamar Hydraulic Hand Dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinem Ayyıldız Çinar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No